CLINICAL TRIAL: NCT03242603
Title: Pilot Study of Anti-GD2 and Expanded, Activated Natural Killer Cell Infusion for Neuroblastoma
Brief Title: Immunotherapy of Neuroblastoma Patients Using a Combination of Anti-GD2 and NK Cells
Acronym: NKEXPGD2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKEXPGD2
Record Dates: First submitted 2017-07-13; First posted 2017-08-08 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2017-06

CONDITIONS: Neuroblastoma Recurrent
Keywords: Relapsed, Refractory, Neuroblastoma; Anti-GD2; Natural Killer (NK) Cells; Immunotherapy
MeSH Terms: conditions — Recurrence; Neuroblastoma

STUDY DESIGN:
Intervention Model Description: To determine the feasibility, safety and effectiveness of anti-GD2 in combination with expanded, activated NK cells in research participants with Neuroblastoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-GD2 in combination with NK cells (Experimental): This is a single arm study. Patients with high risk neuroblastoma who have residual measurable disease will receive a combination of 5 days of anti-GD2 with expanded activated NK cells.
  Interventions: Biological: Anti-GD2 in combination with NK cells

INTERVENTIONS:
Biological: Anti-GD2 in combination with NK cells — Haploidentical donor NK cells will be expanded over 10 days and infused in combination with anti-GD2. Anti-GD2 will be given as daily infusion for 5 days ; D-1, 0,+1, +2 and +3. NK cells will be infused at single dose on day 0. The patient will receive cyclophosphamide 60mg/kg on day -3 and day -2 prior to the NK cell infusion. IL- 2 will be given subcutaneously for 6 doses every alternate day starting on day -1, for NK cell survival.

SUMMARY:
Neuroblastoma is a neoplasm of the sympathetic nervous system which affects mostly children younger than 5 years of age. It is a heterogeneous disease, with nearly 50% of patients presenting with a high-risk phenotype. After standard treatment, the 2-year event-free survival (EFS) for high risk neuroblastoma (EFS) is only about 50%. Immunotherapy with anti-GD2 antibodies has been shown to improve EFS in Children's Oncology Group and SIOPEN trials.

The anti-GD2 antibody mediates neuroblastoma cell killing primarily through antibody-dependent cell-mediated cytotoxicity (ADCC). Natural killer (NK) cells are the main effectors of ADCC. We postulate that infusion of expanded activated NK cells from healthy haploidentical donors along with anti-GD2 antibody will enhance neuroblastoma killing.

DETAILED DESCRIPTION:
Adoptive transfer of haploidentical NK cells has been shown to be safe in clinical trials at NUH. There is experience combining antibody infusion with autologous NK cells in the clinical trial with good safety data.

The proposed trial is a phase I/II study to determine the safety and efficacy of expanded activated haploidentical NK cells in combination with anti-GD2 (ch14.18/CHO). We plan to enrol patients with high risk or relapsed neuroblastoma with evidence of residual disease who are at high risk of recurrence or progression on current treatment.

In the proposed protocol , we plan to infuse NK cells at escalating dose levels to find the optimum dose tolerated by the patients in combination with anti-GD2 (ch14.18/CHO) . There are 3 NK cell dose levels :

Dose level 1 (1 x 10^6/kg) , Dose level 2 (1 x 10^7/kg) , Dose level 3 (1 x 10^8/kg)

If a partial response or stable disease is observed, further infusions of NK cells can be administered. There will be intra- and inter - patient dose escalation.

The donor will be either parent, based on the best NK cell donor as determined by the study team. The donor will be harvested and NK cells expanded prior to infusion into the patient along with anti-GD2 (ch14.18/CHO).

The study aims to study safety and efficacy of a combination of NK cells and anti-GD2 (ch14.18/CHO).

ELIGIBILITY:
Inclusion Criteria:

-

A) Inclusion criteria for activated NK cell Recipient:

1. Age 6 months to 25 years old.
2. Patients with high risk or relapsed neuroblastoma who have measurable residual disease (based on imaging findings with Curie scoring or MIBG or PET imaging criteria) after receiving or has refused to receive standard therapy.

   1. High risk will be defined as stage IV disease with poor response to chemotherapy. Residual disease after surgery or prior to autologous stem cell rescue which is part of Standard of Care. Infants with nMYC amplification will not automatically qualify for the protocol unless they have residual disease after surgery.
   2. Recurrence after completion of standard treatment.
3. Shortening fraction greater than or equal to 25% or Left ventricular ejection fraction (LVEF) greater than or equal to 40%.
4. Glomerular filtration rate greater than or equal to 60 ml/min/1.73 m2.
5. Pulse oximetry greater than or equal to 92% on room air.
6. Direct bilirubin less than or equal to 3.0 mg/dL (50 mmol/L).
7. Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal.
8. Aspartate transaminases (AST) is no more than 2 times the upper limit of normal.
9. Karnofsky or Lansky performance score of greater than or equal to 50.
10. Does not have a current pleural or pericardial effusion.
11. Has a suitable adult family member donor available for NK cell donation.
12. Has recovered from all acute NCI Common Terminology Criteria for Adverse Events (CTCAE) grade II-IV non-hematologic acute toxicities resulting from prior therapy per the judgment of the PI.
13. At least two weeks since receipt of any biological therapy, systemic chemotherapy, and/or radiation therapy.
14. Is not receiving more than the equivalent of prednisone 10 mg daily.
15. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
16. Not lactating.

B) Inclusion criteria for NK cell Donor:

1. First and second degree relative acceptable.
2. 18 years of age or above.
3. Not lactating.
4. Greater than or equal to 3 of 6 HLA match to recipient.
5. .Meets eligibility and suitability criteria for hematopoietic cells donation as per institutional guidelines.
6. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).

Exclusion Criteria:

* Failure to meet any of the above criteria

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
To measure tumor response after infusion of expanded activated haploidentical NK cells with anti-GD2. Response will be assessed as defined by Revised International Neuroblastoma Response Criteria 2017. | 2 years
  Disease status at primary and metastatic soft tissue sites will be assessed using MIBG scans or PET scan as applicable. RECIST and Curie scoring systems will be used to assess response. Metastatic bone disease will be assessed using MIBG or PET scan. Bone marrow will be assessed by histology or flow cytometry. Disease response will be defined as Complete response/remission (CR), Partial response (PR), Minor response, Stable disease (SD), or Progressive disease(PD).

SECONDARY OUTCOMES:
To measure the numbers of infused NK cells in peripheral blood at specific time-points after NK cell infusion | 2 years
  NK cells will be identified by flow cytometry in peripheral blood and their percentages and absolute numbers will be calculated.
To measure cytokine levels in plasma at specific time-points after NK cell infusion | 2 years
  Cytokine panel to assess levels of IL15 serially post lymphodepletion regimen

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kimpo, MD, Principal Investigator — National University Hospital, Singapore; Dario Campana, MD, PhD, Principal Investigator — National University Singapore, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
TBC

REFERENCES:
- [Background] Yu AL, Gilman AL, Ozkaynak MF, London WB, Kreissman SG, Chen HX, Smith M, Anderson B, Villablanca JG, Matthay KK, Shimada H, Grupp SA, Seeger R, Reynolds CP, Buxton A, Reisfeld RA, Gillies SD, Cohn SL, Maris JM, Sondel PM; Children's Oncology Group. Anti-GD2 antibody with GM-CSF, interleukin-2, and isotretinoin for neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1324-34. doi: 10.1056/NEJMoa0911123. PMID 20879881
- [Background] Cho D, Shook DR, Shimasaki N, Chang YH, Fujisaki H, Campana D. Cytotoxicity of activated natural killer cells against pediatric solid tumors. Clin Cancer Res. 2010 Aug 1;16(15):3901-9. doi: 10.1158/1078-0432.CCR-10-0735. Epub 2010 Jun 11. PMID 20542985
- [Background] Tarek N, Le Luduec JB, Gallagher MM, Zheng J, Venstrom JM, Chamberlain E, Modak S, Heller G, Dupont B, Cheung NK, Hsu KC. Unlicensed NK cells target neuroblastoma following anti-GD2 antibody treatment. J Clin Invest. 2012 Sep;122(9):3260-70. doi: 10.1172/JCI62749. Epub 2012 Aug 6. PMID 22863621